CLINICAL TRIAL: NCT04015648
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Zika Virus (ZIKV) Vaccine ChAdOx1 Zika in Healthy Adult Volunteers.
Brief Title: Safety and Immunogenicity of a Candidate ZIKV Vaccine (ZIKA001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIKA001
Record Dates: First submitted 2019-06-04; First posted 2019-07-11 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-11

CONDITIONS: Zika
Keywords: Vaccine
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Volunteers will receive standalone dose of ChAdOx1 Zika 5 x 10^9 vp vaccination intramuscularly.
  Interventions: Biological: ChAdOx1 Zika
- Group 2 (Experimental): Volunteers will receive standalone dose of ChAdOx1 Zika 2.5 x 10^10 vp vaccination intramuscularly.
  Interventions: Biological: ChAdOx1 Zika
- Group 3 (Experimental): Volunteers will receive standalone dose of ChAdOx1 Zika 5 x 10^10 vp vaccination intramuscularly.
  Interventions: Biological: ChAdOx1 Zika

INTERVENTIONS:
Biological: ChAdOx1 Zika — Single dose of ChAdOx1 Zika at different concentrations: 5 x 10^9 vp, 2.5 x 10^10 vp, 5 x 10^10 vp

SUMMARY:
This is a FIH, open-label, dose escalation, phase I clinical trial to assess the safety and immunogenicity of the candidate ChAdOx1 Zika vaccine in healthy volunteers administered intramuscularly.

DETAILED DESCRIPTION:
Volunteers will be recruited and vaccinated at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford. There will be 3 study groups and a total of 24 volunteers will be enrolled. Groups 1-3 will receive ChAdOx1 Zika alone. Staggered enrolment will apply for the first three volunteers within each group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner or access to this medical history electronically (or providing their medical case summaries)
* Women of child-bearing potential agree to practice continuous effective contraception (see below) during the study and test negative for pregnancy on the day(s) of screening and vaccination.
* Agreement to refrain from blood donation during the course of the study
* Agreement to inform study team of any impending vaccinations either before or during participation in the study.
* Agreement to refrain from receipt of any flavivirus vaccine throughout the duration of the study (e.g. investigational or licensed Yellow Fever, Japanese Encephalitis, Tick Borne Encephalitis or Dengue virus vaccines).
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccine, Zika virus vaccine, Dengue virus vaccine).
* Prior receipt of any vaccines administered ≤30 days before enrolment and/or planned receipt of a vaccine ≤30 days after enrolment EXCEPT for protein, RNA (or other non-adenovirus based) COVID-19 vaccinations which may be given within 14 days of the trial vaccine.
* Receipt of recombinant simian adenoviral vaccine prior to enrolment.
* Planned receipt of another adenoviral vectored vaccine (e.g. Oxford/Astrazeneca or Janssen COVID-19 vaccines) within 90 days after the vaccination with the ChAdOx1 Zika
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Any history of anaphylaxis in relation to vaccination.
* History of autoimmune disease.
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Has history of chronic or acute severe neurologic condition. Including: Neurologic and Neuroinflammatory Disorders: ADEM, including site specific variants, Cranial Nerve Disorders (including paralyses/paresis), GBS (including Miller Fisher Syndrome and other variants), Immune-mediated Peripheral Neuropathies and Plexopathies, Optic Neuritis, Multiple Sclerosis, Narcolepsy, Transverse Myelitis, meningitis, or meningoencephalitis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate or access this medical history electronically.
* Seropositivity or cross-reactivity to Zika virus or Dengue virus (serology will be requested at the discretion of the investigator).
* Travel to a Zika virus and/or Dengue virus, endemic region in the 30 days prior to screening, until enrolment and in the first 6 months of the participants enrolment in the study (consult clinical team regarding international travel plans)
* History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism), history of antiphospholipid syndrome, or history of heparin induced thrombocytopenia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ChAdOx1 Zika given as a standalone vaccine at different doses in healthy adult volunteers assessed by the occurrence of solicited adverse events. | Assessment of solicited AEs in the first 7 days post vaccination.
  Occurrence of solicited local and systemic adverse events (i.e: pain, redness, swelling and pruritus at injection site and temperature, feverishness, myalgia, arthralgia, malaise, headache and nausea).
Safety and tolerability of ChAdOx1 Zika given as a standalone vaccine at different doses in healthy adult volunteers assessed by the occurrence of unsolicited adverse events. | Unsolicited AEs to be assessed up to 28 days post vaccination.
  Occurrence of unsolicited local and systemic adverse events
Safety and tolerability of ChAdOx1 Zika given as a standalone vaccine at different doses in healthy adult volunteers assessed by the occurrence of serious adverse events. | SAEs will be collected from enrolment until the end of the follow-up period (i.e. 6 months)
  Occurrence of serious adverse events
Safety and tolerability of ChAdOx1 Zika given as a standalone vaccine at different doses in healthy adult volunteers assessed by the occurrence of laboratory adverse events. | At Day 0 (baseline), day 2, day 7 and day 28 post vaccination
  Occurrence of laboratory adverse events defined as clinically significant changes from baseline. Haematology (Full Blood Count) and Biochemistry (Kidney and Liver Function Tests) will be assessed.

SECONDARY OUTCOMES:
Measures of humoral immunogenicity to the ChAdOx1 ZIKA vaccine | At days 0, 7, 14, 28, 56, 90 and 182 + extended visit days 270 and 360
  ELISA to quantify antibodies to ZIKV protein antigens
Measures of cellular immunogenicity to the ChAdOx1 ZIKA vaccines | At days 0, 7, 14, 28, 56, 90 and 182 + extended visit days 270 and 360
  Ex vivo interferon gamma ELISpot responses to ZIKV protein antigens

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom